CLINICAL TRIAL: NCT01092143
Title: A Randomized, Double Blind, Placebo and Active Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of 6-week Treatment With Oral Doses of 50 mg b.i.d., 200 mg b.i.d., and 400 mg b.i.d. BI 671800 ED in Steroid-naïve Patients With Persistent Asthma
Brief Title: BI 671800 ED in Steroid-naive Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1268.17
Record Dates: First submitted 2010-03-19; First posted 2010-03-24 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — BI 671800; Fluticasone

ARMS (5):
- BI 671800 (low dose) (Experimental): Patients receive BI 671800 (low dose) capsules twice daily
  Interventions: Drug: BI 671800; Drug: Fluticasone propionate placebo
- Fluticasone propionate (Active Comparator): Patients inhale from Fluticasone propionate metered dose inhaler (MDI) twice daily
  Interventions: Drug: Fluticasone propionate; Drug: BI 671800 Placebo
- Placebo (Placebo Comparator): Patients receive placebo capsules twice daily
  Interventions: Drug: Fluticasone propionate placebo; Drug: BI 671800 Placebo
- BI 671800 (medium dose) (Experimental): Patients receive BI 671800 (medium dose) capsules twice daily
  Interventions: Drug: BI 671800; Drug: Fluticasone propionate placebo
- BI 671800 (high dose) (Experimental): Patients receive BI 671800 (high dose) capsules twice daily
  Interventions: Drug: BI 671800; Drug: Fluticasone propionate placebo

INTERVENTIONS:
Drug: BI 671800 — BI 671800
  Arms: BI 671800 (high dose); BI 671800 (low dose); BI 671800 (medium dose)
Drug: Fluticasone propionate placebo — Placebo matching Fluticasone propionate
  Arms: BI 671800 (high dose); BI 671800 (low dose); BI 671800 (medium dose); Placebo
Drug: Fluticasone propionate — Fluticasone propionate
  Arms: Fluticasone propionate
Drug: BI 671800 Placebo — Placebo matching BI 671800
  Arms: Fluticasone propionate; Placebo

SUMMARY:
This is a 6 week study to investigate the effectiveness and safety of BI 671800 ED in patients with asthma who do not take inhaled corticosteroids.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent consistent with ICH-GCP
2. Three month history of reversible (12% with 200 mL) asthma (according to GINA) with following spirometry at randomization: FEV1 60%-85%.
3. No ICS previous 3 months prior to screening.
4. Diagnosis of asthma prior to 40 years.
5. ACQ at least 1.5 at randomization.
6. Male or female, 18 to 65 years.
7. Non-smokers or ex-smokers ( less than 10 pack year history) with negative cotinine screen.
8. Able to perform PFT

Exclusion criteria:

1. Significant diseases other than asthma or allergic rhinitis.
2. Hepatic transaminases or total bilirubin greater than 1.5 ULN.
3. Hospitalizations for asthma or asthma related intubation within 3 months.
4. Uncontrolled asthma.
5. Respiratory tract infection or exacerbation within 4 weeks.
6. FEV1 less than 40%, more than 12 puffs of SABA on more than two consecutive days or asthma exacerbation during the run-in period.
7. Participation in another interventional study.
8. Pregnant or nursing women.
9. Women of child bearing potential nor using appropriate methods of birth control as defined by protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2010-03-18 (Actual); Primary Completion 2011-03-26 (Actual); Study Completion 2011-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (92):
- United States (40):
  - 1268.17.01043 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1268.17.01009 Boehringer Ingelheim Investigational Site, Cypress, California
  - 1268.17.01006 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1268.17.01040 Boehringer Ingelheim Investigational Site, Palmdale, California
  - 1268.17.01024 Boehringer Ingelheim Investigational Site, San Jose, California
  - 1268.17.01003 Boehringer Ingelheim Investigational Site, Stockton, California
  - 1268.17.01015 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1268.17.01001 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1268.17.01016 Boehringer Ingelheim Investigational Site, Lakewood, Colorado
  - 1268.17.01033 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1268.17.01045 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1268.17.01036 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 1268.17.01025 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 1268.17.01005 Boehringer Ingelheim Investigational Site, Iowa City, Iowa
  - 1268.17.01034 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1268.17.01014 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1268.17.01030 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1268.17.01027 Boehringer Ingelheim Investigational Site, Novi, Michigan
  - 1268.17.01032 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1268.17.01010 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1268.17.01037 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1268.17.01022 Boehringer Ingelheim Investigational Site, Bozeman, Montana
  - 1268.17.01008 Boehringer Ingelheim Investigational Site, Bellevue, Nebraska
  - 1268.17.01011 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1268.17.01004 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1268.17.01038 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1268.17.01042 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1268.17.01007 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1268.17.01031 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1268.17.01039 Boehringer Ingelheim Investigational Site, Fort Mill, South Carolina
  - 1268.17.01026 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1268.17.01029 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1268.17.01049 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1268.17.01019 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1268.17.01012 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 1268.17.01023 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1268.17.01048 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1268.17.01028 Boehringer Ingelheim Investigational Site, New Braunfels, Texas
  - 1268.17.01035 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1268.17.01047 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- 1268.17.61001 Boehringer Ingelheim Investigational Site, Adelaide, South Australia, Australia
- Canada (8):
  - 1268.17.02015 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1268.17.02012 Boehringer Ingelheim Investigational Site, Hawkesbury, Ontario
  - 1268.17.02010 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1268.17.02014 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1268.17.02003 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1268.17.02013 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1268.17.02001 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1268.17.02004 Boehringer Ingelheim Investigational Site, Québec, Quebec
- Colombia (3):
  - 1268.17.57003 Boehringer Ingelheim Investigational Site, Bogotá
  - 1268.17.57004 Boehringer Ingelheim Investigational Site, Bogotá
  - 1268.17.57002 Boehringer Ingelheim Investigational Site, Medellín
- Mexico (4):
  - 1268.17.52002 Boehringer Ingelheim Investigational Site, Cuernavaca
  - 1268.17.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1268.17.52004 Boehringer Ingelheim Investigational Site, Toriello Guerra
  - 1268.17.52003 Boehringer Ingelheim Investigational Site, Zona Río
- New Zealand (3):
  - 1268.17.64001 Boehringer Ingelheim Investigational Site, Christchurch
  - 1268.17.64003 Boehringer Ingelheim Investigational Site, Greenlane East Auckland
  - 1268.17.64002 Boehringer Ingelheim Investigational Site, Newtown Wellington NZ
- Peru (6):
  - 1268.17.51003 Boehringer Ingelheim Investigational Site, Jesús María
  - 1268.17.51002 Boehringer Ingelheim Investigational Site, Lima
  - 1268.17.51006 Boehringer Ingelheim Investigational Site, San Borja
  - 1268.17.51004 Boehringer Ingelheim Investigational Site, San Isidro
  - 1268.17.51005 Boehringer Ingelheim Investigational Site, Santiago de Surco
  - 1268.17.51001 Boehringer Ingelheim Investigational Site, Urb. Ingeniería
- Philippines (7):
  - 1268.17.63007 Boehringer Ingelheim Investigational Site, Caloocan
  - 1268.17.63002 Boehringer Ingelheim Investigational Site, Manila
  - 1268.17.63001 Boehringer Ingelheim Investigational Site, Quezon City
  - 1268.17.63003 Boehringer Ingelheim Investigational Site, Quezon City
  - 1268.17.63004 Boehringer Ingelheim Investigational Site, Quezon City
  - 1268.17.63005 Boehringer Ingelheim Investigational Site, Quezon City
  - 1268.17.63006 Boehringer Ingelheim Investigational Site, Quezon City
- South Korea (8):
  - 1268.17.82007 Boehringer Ingelheim Investigational Site, Cheongju-si
  - 1268.17.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.17.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.17.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.17.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.17.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.17.82003 Boehringer Ingelheim Investigational Site, Suwon
  - 1268.17.82008 Boehringer Ingelheim Investigational Site, Wŏnju
- Taiwan (12):
  - 1268.17.86210 Boehringer Ingelheim Investigational Site, Chiayi City
  - 1268.17.86211 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1268.17.86207 Boehringer Ingelheim Investigational Site, Taichung
  - 1268.17.86208 Boehringer Ingelheim Investigational Site, Taichung
  - 1268.17.86209 Boehringer Ingelheim Investigational Site, Taichung
  - 1268.17.86201 Boehringer Ingelheim Investigational Site, Taipei
  - 1268.17.86202 Boehringer Ingelheim Investigational Site, Taipei
  - 1268.17.86203 Boehringer Ingelheim Investigational Site, Taipei
  - 1268.17.86204 Boehringer Ingelheim Investigational Site, Taipei
  - 1268.17.86205 Boehringer Ingelheim Investigational Site, Taipei
  - 1268.17.86206 Boehringer Ingelheim Investigational Site, Taipei
  - 1268.17.86200 Boehringer Ingelheim Investigational Site, Taoyuan

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIa multi-centre, multi-national, randomized, double-blind, placebo-controlled, parallel group, double-dummy study investigating the efficacy, safety and tolerability of BI 671800 ED (50, 200 and 400 mg b.i.d.) compared to fluticasone propionate 110 mcg 2 puffs b.i.d. and placebo in symptomatic steroid-naïve asthma patients.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all subjects as required.
Groups:
- Placebo: Daily treatment with 4 oral capsules of Placebo and 2 puffs Placebo metered dose inhaler (MDI) 110 microgram (mcg) in the morning and 4 oral capsules of Placebo and 2 puffs Placebo MDI 110 mcg in the evening, for a total treatment period of 6 weeks.
- BI 671800 50 mg Bid: Daily treatment with 2 oral capsules of 25 milligram (mg) BI 671800 Ethylenediamine (ED), 2 oral capsules of Placebo and 2 puffs Placebo metered dose inhaler (MDI) 110 microgram (mcg) in the morning and 2 oral capsules of 25 mg BI 671800 ED, 2 oral capsules of Placebo and 2 puffs Placebo MDI 110 mcg in the evening, for a total treatment period of 6 weeks.
- BI 671800 200 mg Bid: Daily treatment with oral 2 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED), 2 oral capsules of Placebo and 2 puffs Placebo metered dose inhaler (MDI) 110 microgram (mcg) in the morning and 2 oral capsules of 100 mg BI 671800 ED, 2 oral capsules of Placebo and 2 puffs Placebo MDI 110 mcg in the evening, for a total treatment period of 6 weeks.
- BI 671800 400 mg Bid: Daily treatment with 4 oral capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) and 2 puffs Placebo metered dose inhaler (MDI) 110 microgram (mcg) in the morning and 4 oral capsules of 100 mg BI 671800 ED and 2 puffs Placebo MDI 110 mcg in the evening, for a total treatment period of 6 weeks.
- Fluticasone 220 mcg Bid: Daily treatment with 4 oral capsules of Placebo and 2 puffs Fluticasone propionate metered dose inhaler (MDI) 110 microgram (mcg) in the morning and 4 oral capsules of Placebo and 2 puffs Fluticasone propionate MDI 110 mcg in the evening, for a total treatment period of 6 weeks.
Period: Overall Study
Arm/Group | Placebo | BI 671800 50 mg Bid | BI 671800 200 mg Bid | BI 671800 400 mg Bid | Fluticasone 220 mcg Bid
Started | 78 | 77 | 84 | 79 | 71
Treated | 78 | 77 | 83 | 79 | 71
Completed | 63 | 70 | 80 | 72 | 63
Not Completed | 15 | 7 | 4 | 7 | 8
Not completed — Adverse Event | 10 | 5 | 1 | 4 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Consent withdrawn | 2 | 1 | 0 | 1 | 3
Not completed — Not treated | 0 | 0 | 1 | 0 | 0
Not completed — did not reversibility criteria | 0 | 0 | 1 | 0 | 0
Not completed — Increased Albuterol use for >2 days | 0 | 1 | 0 | 0 | 0
Not completed — Ineligible patient | 1 | 0 | 0 | 0 | 0
Not completed — Drop in FEV1 at visit 9 | 1 | 0 | 0 | 0 | 0
Not completed — Patient travel | 0 | 0 | 0 | 0 | 1
Not completed — Non compliance with study medication | 0 | 0 | 0 | 0 | 1
Not completed — Randomized by mistake | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All randomized patients who received at least one dose of treatment, the treated set was used in the safety analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 671800 50 mg Bid | BI 671800 200 mg Bid | BI 671800 400 mg Bid | Fluticasone 220 mcg Bid | Total
Number analyzed (Participants) | 78 | 77 | 83 | 79 | 71 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.99) | 39.1 (11.53) | 35.1 (11.09) | 37.5 (12.23) | 39.4 (12.20) | 37.4 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 42 | 43 | 36 | 199
  Male | 41 | 36 | 41 | 36 | 35 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 17 | 20 | 20 | 23 | 100
  Not Hispanic or Latino | 56 | 58 | 60 | 57 | 45 | 276
  Unknown or Not Reported | 2 | 2 | 3 | 2 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 10 | 12 | 13 | 11 | 57
  Asian | 13 | 13 | 19 | 13 | 13 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 0 | 2
  Black or African American | 12 | 11 | 9 | 10 | 5 | 47
  White | 42 | 42 | 43 | 42 | 42 | 211
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Percentage of predicted forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: Percentage of predicted FEV1] | 70.811 (8.6801) | 68.812 (10.6335) | 72.626 (9.9901) | 71.646 (7.4747) | 70.481 (9.7577) | 70.904 (9.4014)

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) % Predicted Trough Change From Baseline (Mean Observed in the 2 Weeks Prior to Treatment) After Six Weeks of Treatment
Description: Forced expiratory volume in one second (FEV1) % predicted trough change from baseline (mean observed in the 2 weeks prior to treatment) after 6 weeks of treatment, where trough FEV1 % predicted was defined as the mean of the FEV1 % predicted trough values at 25 minutes and 10 minutes prior to dosing on clinic visit.
  MMRM in the statistical test comments is mixed effects model with repeated measures.
Time Frame: Measurements at baseline (mean observed in the 2 weeks prior to treatment) and at week 6 of treatment.
Population: Statistical analysis was performed on the Full Analysis Set (FAS): Randomized patients who received at least one dose of treatment and had both baseline and at least one post-baseline measurement at or before 6 weeks for the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: FEV1 percent predicted
Arm/Group | Placebo | BI 671800 50 mg Bid | BI 671800 200 mg Bid | BI 671800 400 mg Bid | Fluticasone 220 mcg Bid
Number analyzed (Participants) | 63 | 69 | 81 | 71 | 63
FEV1 percent predicted | -2.010 (1.187) | 1.073 (1.144) | 1.580 (1.074) | 1.967 (1.133) | 6.610 (1.194)
Statistical Analysis 1: Comparison: Placebo vs BI 671800 50 mg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with BI 671800 50 mg b.i.d. compared with those treated with placebo, after 6 weeks; Test type: Superiority; p = 0.0311, Mixed Models Analysis — α=0.025 one-sided; MMRM with baseline, treatment, day, treatment by day interaction and baseline by day interaction as fixed effects and patient as a random effect; Adjusted mean treatment differences = 3.083, 95% CI 2-sided [-0.157 to 6.323], Standard Deviation 1.650
Statistical Analysis 2: Comparison: Placebo vs BI 671800 200 mg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with BI 671800 200 mg b.i.d. compared with those treated with placebo, after 6 weeks; Test type: Superiority; p = 0.0126, Mixed Models Analysis — α=0.025 one-sided; MMRM with baseline, treatment, day, trea; Adjusted mean treatment differences = 3.589, 95% CI 2-sided [0.447 to 6.732], Standard Deviation 1.600
Statistical Analysis 3: Comparison: Placebo vs BI 671800 400 mg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with BI 671800 400 mg b.i.d. compared with those treated with placebo, after 6 weeks; Test type: Superiority; p = 0.0078, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 3.977, 95% CI 2-sided [0.756 to 7.197], Standard Deviation 1.640
Statistical Analysis 4: Comparison: Placebo vs Fluticasone 220 mcg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with fluticasone propionate 110 mcg 2 puffs b.i.d. compared with those treated with placebo, after 6 weeks; Test type: Other; p < .0001, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 8.619, 95% CI 2-sided [5.312 to 11.927], Standard Deviation 1.684
Statistical Analysis 5: Comparison: BI 671800 50 mg Bid vs Fluticasone 220 mcg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with BI 671800 50 mg b.i.d. compared with those treated with fluticasone propionate 220 mcg b.i.d., after 6 weeks; Test type: Superiority; p = 0.9996, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -5.536, 95% CI 2-sided [-8.783 to -2.290], Standard Deviation 1.653
Statistical Analysis 6: Comparison: BI 671800 200 mg Bid vs Fluticasone 220 mcg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with BI 671800 200 mg b.i.d. compared with those treated with fluticasone propionate 220mcg b.i.d., after 6 weeks; Test type: Superiority; p = 0.9991, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -5.030, 95% CI 2-sided [-8.185 to -1.875], Standard Deviation 1.606
Statistical Analysis 7: Comparison: BI 671800 400 mg Bid vs Fluticasone 220 mcg Bid; Superiority in mean trough FEV1 % predicted change from baseline in patients treated with BI 671800 400 mg b.i.d. compared with those treated with fluticasone propionate 220 mcg b.i.d., after 6 weeks; Test type: Superiority; p = 0.9975, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -4.643, 95% CI 2-sided [-7.877 to -1.408], Standard Deviation 1.647

2. Secondary Outcome: Asthma Control Questionnaire (ACQ) Mean Score Change From Baseline After Six Weeks of Treatment
Description: Asthma Control Questionnaire (ACQ) mean score change from baseline (mean ACQ score obtained at Week 0) after six weeks of treatment.
  The Asthma Control Questionnaire (ACQ) is a patient-reported outcome questionnaire containing 7 items. The items are equally weighted and the ACQ score is the mean of the 7 items and therefore between 0 (well controlled) and 6 (extremely poorly controlled) These questions based on recall of the previous 7 days comprise breathlessness, nocturnal waking, symptoms on waking, activity limitation, wheeze, frequency of short-acting beta-adrenergic (SABA) use, and categorized pre-bronchodilator FEV1% predicted.
Time Frame: Measurements at baseline (mean ACQ score obtained at Week 0) and at week 6 of treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | BI 671800 50 mg Bid | BI 671800 200 mg Bid | BI 671800 400 mg Bid | Fluticasone 220 mcg Bid
Number analyzed (Participants) | 64 | 69 | 81 | 71 | 63
Score on a scale | -0.616 (0.081) | -0.543 (0.078) | -0.696 (0.074) | -0.677 (0.078) | -0.949 (0.082)
Statistical Analysis 1: Comparison: Placebo vs BI 671800 50 mg Bid; Test type: Superiority; p = 0.7413, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 0.073, 95% CI 2-sided [-0.149 to 0.295], Standard Deviation 0.113
Statistical Analysis 2: Comparison: Placebo vs BI 671800 200 mg Bid; Test type: Superiority; p = 0.2335, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -0.080, 95% CI 2-sided [-0.296 to 0.136], Standard Deviation 0.110
Statistical Analysis 3: Comparison: Placebo vs BI 671800 400 mg Bid; Test type: Superiority; p = 0.2933, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -0.061, 95% CI 2-sided [-0.282 to 0.160], Standard Deviation 0.113
Statistical Analysis 4: Comparison: Placebo vs Fluticasone 220 mcg Bid; Test type: Superiority; p = 0.0021, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -0.333, 95% CI 2-sided [-0.561 to -0.105], Standard Deviation 0.116
Statistical Analysis 5: Comparison: BI 671800 50 mg Bid vs Fluticasone 220 mcg Bid; Test type: Superiority; p = 0.9998, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 0.406, 95% CI 2-sided [0.183 to 0.630], Standard Deviation 0.114
Statistical Analysis 6: Comparison: BI 671800 200 mg Bid vs Fluticasone 220 mcg Bid; Test type: Superiority; p = 0.9890, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 0.253, 95% CI 2-sided [0.037 to 0.470], Standard Deviation 0.110
Statistical Analysis 7: Comparison: BI 671800 400 mg Bid vs Fluticasone 220 mcg Bid; Test type: Superiority; p = 0.9918, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 0.272, 95% CI 2-sided [0.050 to 0.494], Standard Deviation 0.113

ADVERSE EVENTS:
Time Frame: Adverse Events: Day of the first dose till the day of the last dose + 5 days residual effect period, up to 61 days. All-Cause Mortality: Day of the first dose till the day of the last dose + 2 weeks follow up, up to 70 days.
Description: Treated Set (TS): All randomized patients who received at least one dose of treatment, the treated set was used in the safety analysis.
Arm/Group | Placebo | BI 671800 50 mg Bid | BI 671800 200 mg Bid | BI 671800 400 mg Bid | Fluticasone 220 mcg Bid
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/77 | 0/83 | 0/79 | 0/71
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/77 | 0/83 | 1/79 | 0/71
Other Adverse Events (participants affected / at risk) | 14/78 | 15/77 | 9/83 | 14/79 | 11/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=78) | BI 671800 50 mg Bid (N=77) | BI 671800 200 mg Bid (N=83) | BI 671800 400 mg Bid (N=79) | Fluticasone 220 mcg Bid (N=71)
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=78) | BI 671800 50 mg Bid (N=77) | BI 671800 200 mg Bid (N=83) | BI 671800 400 mg Bid (N=79) | Fluticasone 220 mcg Bid (N=71)
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 5 | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 3 | 5 | 2
Headache (Nervous system disorders) | 0 | 4 | 3 | 4 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights